CLINICAL TRIAL: NCT02738814
Title: Clinical Study on the Effects of Propofol for Treatment on Emergence Agitation After Sevoflurane Anesthesia in Pediatric Strabismus Surgery
Brief Title: Propofol for Treatment on Emergence Agitation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sangjae Park, resident, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ED15301
Record Dates: First submitted 2016-03-01; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Child; Anesthesia Morbidity
Keywords: emergence agitation; emergence delirium; PAED scale; The Modified Aldrete Scoring System; treatment; pediatric; sevoflurane
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAED > 13 (Experimental): When severe emergence agitation(PAED is 14 or more) is occured, Pharmacologic treatment of emergence agitation relies on the administration of IV propofol 0.8 or 1 mg/kg.
  Interventions: Drug: propofol
- PAED < 14 (No Intervention): Caregivers must first try to reassure patients.

INTERVENTIONS:
Drug: propofol — When severe emergence agitation(PAED > 13) is occurred, Pharmacologic treatment of emergence agitation relies on the administration of IV propofol 0.8 or 1 mg/kg.
  Other Names: fresofol MCT 1%
  Arms: PAED > 13

SUMMARY:
This study aimed to verify the effects of propofol for treatment on emergence agitation (EA) after sevoflurane anesthesia in pediatric strabismus surgery.

DETAILED DESCRIPTION:
Sevoflurane with rapid anesthetic induction and emergence, hemodynamic stability, and nonirritating airway properties, has acquired widespread acceptance in children. However, sevoflurane has been reported to be associated with emergence agitation in children, with a reported incidence of up to 80%. In severe case, it cause injury to the child or to the surgical site and lead to the accidental removal of surgical dressings and intravenous catheters. In case of intense agitation with high risk of self-injury, pharmacologic intervention seems reasonable. Pharmacologic treatment of emergence agitation relies on the administration of IV sedative agents (IV midazolam 0.1 mg/kg12 or propofol 0.5 or 1 mg/kg) or opioid agents (IV fentanyl 1 or 2 mcg/kg). However, these treatments are empirical and were extrapolated from pharmacologic preventive studies performed at the end of surgery or from personal experience. To the investigators knowledge, there is no risk of recurrence of EA after a first episode. Consequently, EA is not per se a factor of increased duration of PACU (post-anaesthesia care unit ) stay, but sedative or opioid agents administered postoperatively to alleviate it might prolong this stay.

Therefore, the investigators design a study to confirm statistically effect of propofol for treatment on emergence agitation after sevoflurane anesthesia in pediatric strabismus surgery through PAED scale. Furthermore duration of PACU stay is checked after propofol administration.

ELIGIBILITY:
Inclusion Criteria:

* ASA (american society of anesthesiologists) physical status patients, aged 3-10yr, presenting for elective strabismus surgery.

Exclusion Criteria:

* Refusal by parents, neurologic disease, developmental delay, history of any previous surgery, American society of Anesthesiologists physical status score of III or IV, and airway disease

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of Emergent Adverse Events [Safety and Tolerability] | From just after extubation until the discharge from PACU, assessed up to 2 hours.
  After anesthetic emergence, investigator, nurse and attending anesthesiologist check the PAED scale every 5min, up to 2 hours until discharge from PACU. If checked PAED scale is 14 or more, attending anesthesiologist administers 1% propofol 0.8~1.0mg/kg(sedative dose). Then they check PAED scale every 5min after the arousal from sedative state until the discharge from PACU.

SECONDARY OUTCOMES:
Duration of PACU stay | From the arrival of the PACU to discharge from the PACU, assessed an average of 1hour
  The investigator check the duration of PACU stay, defined as the interval from the time of arrival of PACU to the time of discharge from PACU, if sadisfacted to discharge criteria score(from Aldrete JA. J Clin Anesth 1995; 7:89-91), a score 9 or more is required for discharge.

CONTACTS AND LOCATIONS:
Overall Officials: SeungZhoo Yoon, M.D.PhD., Study Director — Department of Anesthesiology and Pain medicine. Korea universicy medical center.
Locations (1):
- Korea University Medical Center, Anam hospital, Seoul, Seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu GS, Yoon SZ, Choi YJ, Shin HW, Kim JH. Postoperative propofol bolus treatment did not affect recovery time in patients with emergence agitation after sevoflurane anesthesia in pediatric patients undergoing strabismus surgery: Prospective nonrandomized case-control study. Medicine (Baltimore). 2022 Jul 15;101(28):e29521. doi: 10.1097/MD.0000000000029521. PMID 35838993